CLINICAL TRIAL: NCT03830281
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Humalog in Adults With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion
Brief Title: A Study Comparing LY900014 to Insulin Lispro (Humalog) in Adults With Type 1 Diabetes Using Insulin Pump Therapy
Acronym: PRONTO-Pump-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16315; I8B-MC-ITRO (Other: Eli Lilly and Company); 2015-005358-36 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin Lispro (Humalog) (Active Comparator): Participants received individual dose of 100 U/mL insulin lispro (Humalog) by CSII; where mealtime boluses were delivered 0 to 2 minutes prior to the start of each meal, with basal infusion rates 24 hours/day, and correction boluses as necessary.
  Interventions: Drug: Insulin Lispro
- Ultra-Rapid Lispro (Experimental): Participants received individual dose of 100 units per milliliter (U/mL) ultra rapid lispro by continuous subcutaneous insulin infusion (CSII); where mealtime boluses were delivered 0 to 2 minutes prior to the start of each meal, with basal infusion rates 24 hours/day, and correction boluses as necessary.
  Interventions: Drug: Ultra-Rapid Lispro

INTERVENTIONS:
Drug: Ultra-Rapid Lispro — Administered SC
  Other Names: LY900014; Insulin lispro
  Arms: Ultra-Rapid Lispro
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro (Humalog)

SUMMARY:
The reason for this study is to compare the study drug LY900014 to insulin lispro (Humalog) when both are used in insulin pump therapy in adults with type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with T1D and continuously using insulin for at least 1 year
* Have been using CSII therapy for a minimum of 6 months
* Currently treated with <100 Units of one of following rapid-acting analog insulin via CSII for at least the past 30 days: insulin lispro U-100, insulin aspart, fast-acting insulin aspart, insulin glulisine
* Must be using a MiniMed 530G (US), Paradigm Revel (US), or MiniMed 630G (US and Canada), MiniMed 640G or Paradigm Veo (select countries outside the US), insulin pump for at least the past 90 days

Exclusion Criteria:

* Have hypoglycemia unawareness
* Have had more than 1 episode of severe hypoglycemia within 6 months prior to screening
* Have had more than 1 emergency room visit or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis) within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (82):
- United States (31):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Research, Fresno, California
  - Marin Endocrine Associates, Greenbrae, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - University Clinical Investigators, Inc., Tustin, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - ALL Medical Research, LLC, Cooper City, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Metabolic Research Institute Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - East West Medical Institute, Honolulu, Hawaii
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Northwestern Feinberg School of Medicine, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Iderc, P.L.C., West Des Moines, Iowa
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Physicians East, Greenville, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Texas Diabetes and Endocrinology-Austin South, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Texas Diabetes and Endocrinology, P.A., Round Rock, Texas
  - Private: Dr. Larry Stonesifer, Federal Way, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
- Australia (5):
  - The AIM Centre, Merewether, New South Wales
  - GP Plus Marion, Oaklands Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Barwon Health - The Geelong Hospital, Geelong, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Austria (4):
  - Universitätsklinikum Graz, Graz, Styria
  - VIVIT Institut am LKH Feldkirch, Feldkirch, Vorarlberg
  - Universitätsklinikum Salzburg, Salzburg
  - KA Rudolfstiftung, Vienna
- Canada (6):
  - LMC Endocrinology Centres Ltd., Barrie, Ontario
  - LMC Endocrinology Centres Ltd., Concord, Ontario
  - LMC Endocrinology Centres, Oakville, Ontario
  - LMC Endocrinology Centres Ltd., Toronto, Ontario
  - IRCM, Montreal, Quebec
  - LMC Endocrinology Centres Ltd., Saint-Laurent, Quebec
- France (6):
  - CHU Toulouse Hopital de Rangueil, Toulouse, Cedex 9
  - Clinique Hotel Dieu, Le Creusot
  - Centre hospitalier universitaire Lapeyronie, Montpellier
  - Hopital Cochin, Paris
  - Hôpital de HautePierre, Strasbourg
  - Groupe hospitalier mutualiste Les Portes du sud, Vénissieux
- Germany (8):
  - Arztpraxis Dr. Cornelia Marck, Pohlheim, Hesse
  - Institut für Diabetesforschung Münster GmbH, Münster, North Rhine-Westphalia
  - Praxis Dr. Kempe - Dr. Stemler, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Schwerpunktpraxis Diabetes, Saint Ingbert-Oberwürzbach, Saarland
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetespraxis Prenzlauer Allee, Berlin
  - Diabetologische Schwerpunktpraxis B. Scholz/Dr. B. Paschen, Hamburg
  - Gemeinschaftspraxis für innere Medizin und Diabetologie, Hamburg
- Hungary (4):
  - Budai Irgalmasrendi Korhaz, Budapest
  - ClinDiab Kft., Budapest
  - UNO Medical Trials Kft., Budapest
  - TRANTOR 99 Bt., Budapest
- Israel (5):
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Schneider Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (5):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale San Giovanni di Dio, Olbia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Dip.to Med. Sperimentale -Polic.Umberto I -Univ. La Sapienza, Roma
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón, PR
  - Centro de Endocrinologia Alcantara Gonzalez, Lomas Verdes
- Spain (6):
  - Corporació Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study Comparing LY900014 to Insulin Lispro in Adults With Type 1 Diabetes Using Insulin Pump Therapy — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/ITRO#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The purpose of the lead-in period was to assess basal rates and bolus calculator settings and adjust if needed prior to randomization. Participants (Pts) were then randomized to insulin lispro (Humalog) or ultra-rapid lispro as both basal and bolus insulin and delivered bolus doses 0 to 2 minutes prior to each meal (pre-meal).
Groups:
- Insulin Lispro (Humalog): Participants received individual dose of 100 units per milliliter (U/mL) insulin lispro (Humalog) by continuous subcutaneous insulin infusion (CSII); where mealtime boluses were delivered 0 to 2 minutes prior to the start of each meal, with basal infusion rates 24 hours/day, and correction boluses as necessary.
- Ultra-Rapid Lispro: Participants received individual dose of 100 U/mL ultra rapid lispro by CSII; where mealtime boluses were delivered 0 to 2 minutes prior to the start of each meal, with basal infusion rates 24 hours/day, and correction boluses as necessary.
Period: Lead-in Period (2 Weeks)
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Started | 471 | 0
Completed | 432 | 0
Not Completed | 39 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Not Met Eligibility Criteria | 6 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 29 | 0
Period: Treatment Period (16 Weeks)
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Started | 217 (Pts who completed lead-in period randomized to Humalog or Ultra-Rapid Lispro in treatment period.) | 215 (Pts who completed lead-in period randomized to Humalog or Ultra-Rapid Lispro in treatment period.)
Completed | 205 | 198
Not Completed | 12 | 17
Not completed — Adverse Event | 1 | 7
Not completed — Lost to Follow-up | 4 | 3
Not completed — Sponsor Decision | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro | Total
Number analyzed (Participants) | 217 | 215 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (14.9) | 48.2 (15.4) | 46.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 120 | 239
  Male | 98 | 95 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Not Hispanic or Latino | 180 | 178 | 358
  Unknown or Not Reported | 20 | 19 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 7 | 13
  White | 207 | 202 | 409
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 11 | 22
  Puerto Rico | 2 | 3 | 5
  Austria | 8 | 8 | 16
  Hungary | 24 | 24 | 48
  United States | 86 | 84 | 170
  Italy | 9 | 9 | 18
  Israel | 22 | 19 | 41
  Australia | 15 | 15 | 30
  France | 7 | 7 | 14
  Germany | 17 | 19 | 36
  Spain | 16 | 16 | 32
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 7.54 (0.58) | 7.56 (0.59) | 7.55 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) Efficacy Estimand at Week 16
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates: Baseline + Pooled Country + Personal continuous glucose Monitor (CGM) or Flash glucose monitor (FGM) use during study flag + Treatment + Time + Treatment*Time (Type III sum of squares). The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 207 | 191
Percentage of HbA1c | -0.09 (0.030) | -0.06 (0.031)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs Ultra-Rapid Lispro; Test type: Non-Inferiority — Noninferiority margin = 0.4% for HbA1c; p = 0.565, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.06 to 0.11]

2. Secondary Outcome: Change From Baseline in 1-hour Postprandial Glucose (PPG) During Mixed-Meal Tolerance Test (MMTT) Efficacy Estimand at Week 16
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 1-hour timepoint after the start of meal minus fasting serum glucose. Least Squares (LS) mean was determined by analysis of variance (ANCOVA) model with independent variables: Baseline + Pooled Country + Hemoglobin A1C Stratum + Personal CGM/FGM use during study Flag + Treatment (Type III sum of squares).The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline 1-hour PPG data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 193 | 182
milligrams per deciliter (mg/dL) | -2.2 (5.02) | -26.3 (5.33)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs Ultra-Rapid Lispro; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -24.1, 95% CI 2-sided [-36.0 to -12.2]

3. Secondary Outcome: Change From Baseline in 2-hour PPG During MMTT Efficacy Estimand at Week 16
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 2-hour timepoint after the start of meal minus fasting serum glucose. Least Squares (LS) mean was determined by analysis of variance (ANCOVA) model with independent variables: Baseline + Pooled Country + Hemoglobin A1C Stratum + Personal CGM/FGM use during study Flag + Treatment (Type III sum of squares).The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline 2-hour PPG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 192 | 183
mg/dL | -4.2 (6.27) | -32.0 (6.59)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs Ultra-Rapid Lispro; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -27.8, 95% CI 2-sided [-42.6 to -13.0]

4. Secondary Outcome: Percentage of Time With Sensor Glucose Values Between 70 and 180 mg/dL Efficacy Estimand at Week 16
Description: Percentage of time with sensor glucose values between 70 and 180 mg/dL using continuous glucose monitoring (CGM). Least square (LS) mean difference will provided for CGM data normalized to a 24hrs period. Daytime: 0600 hours to midnight (06:00:00-23:59:59 on the 24-hour clock). Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates: Baseline + Pooled Country + Hemoglobin A1C Stratum + Personal continuous glucose Monitor (CGM) or Flash glucose monitor (FGM) use during study flag + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Week 16
Population: All randomized participants with non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 181 | 172
percentage of time
  Daytime | 58.6 (0.75) | 59.3 (0.77)
  24-Hour: number analyzed (Participants) | 181 | 171
  24-Hour | 57.5 (0.76) | 57.9 (0.79)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs Ultra-Rapid Lispro; Statistical analysis during daytime is reported; Test type: Superiority; p = 0.532, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-1.4 to 2.8]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs Ultra-Rapid Lispro; Statistical analysis during 24-hour period is reported; Test type: Superiority; p = 0.738, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-1.8 to 2.5]

5. Secondary Outcome: Rate of Severe Hypoglycemia at Week 16
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. During these episodes, the participant has an altered mental status and cannot assist in his or her own care, or may be semiconscious or unconscious, or experience coma with or without seizures, and may require parenteral therapy. Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within a treatment group *36525.
Time Frame: Baseline through Week 16
Population: All randomized participants with evaluable hypoglycemic data.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 217 | 214
Events per 100 participant years | 2.95 | 6.36

6. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemia at Week 16
Description: Documented symptomatic hypoglycemia is an event during which typical symptoms of hypoglycemia are accompanied by blood glucose (BG) of <54 mg/dL [3.0 millimole per liter (mmol/L)]. The rate of documented symptomatic hypoglycemia was estimated by negative binomial model: number of episodes = treatment with log (treatment exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Week 16
Population: All randomized participants with evaluable hypoglycemic data.
Measure: Least Squares Mean (Standard Error); unit: Events per participant per year
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 217 | 214
Events per participant per year | 30.7 (2.48) | 24.6 (1.88)

7. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG) at Week 16
Description: 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. 1,5-AG accurately predicts rapid changes in glycemia and is tightly associated with glucose fluctuations and postprandial glucose. LS Mean was calculated using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (Pooled Country + Hemoglobin A1C Stratum + Personal continuous glucose Monitor (CGM) or Flash glucose monitor (FGM) use during study flag), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The analysis included data collected prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline 1,5-AG data.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 202 | 185
milligram per liter (mg/L) | 0.16 (0.116) | 0.11 (0.121)

8. Secondary Outcome: Change From Baseline in 10-Point Self-Monitoring Blood Glucose (SMBG) Values at Week 16
Description: SMBG 10-point profiles were measured at fasting, 1-hour post morning meal, 2-hours post morning meal, pre midday meal, 1-hour post midday meal, 2-hours post midday meal, pre evening meal, 1-hour post evening meal, 2-hours post evening meal, and bedtime. LS Mean was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, HbA1c stratum : less than or equal to (≤)7.5%, greater than (>)7.5% and participant's personal CGM or FGM use during the study), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The efficacy estimand included participant data when baseline and at least one post-baseline measurement prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 195 | 178
mg/dL
  Morning Premeal | 0.2 (2.76) | 0.5 (2.89)
  Morning 1-hour Postmeal: number analyzed (Participants) | 189 | 172
  Morning 1-hour Postmeal | -3.1 (3.15) | -12.9 (3.31)
  Morning 2-hour Postmeal: number analyzed (Participants) | 192 | 172
  Morning 2-hour Postmeal | -2.7 (3.04) | -2.9 (3.21)
  Midday Premeal: number analyzed (Participants) | 195 | 175
  Midday Premeal | -0.6 (2.82) | 4.9 (2.98)
  Midday 1-hour Postmeal: number analyzed (Participants) | 188 | 166
  Midday 1-hour Postmeal | -4.2 (2.85) | -6.3 (3.03)
  Midday 2-hour Postmeal: number analyzed (Participants) | 191 | 171
  Midday 2-hour Postmeal | -0.2 (3.14) | 4.4 (3.31)
  Evening Premeal: number analyzed (Participants) | 193 | 178
  Evening Premeal | 3.8 (3.28) | 17.5 (3.41)
  Evening 1-hour Postmeal: number analyzed (Participants) | 189 | 167
  Evening 1-hour Postmeal | 2.6 (3.21) | 8.6 (3.41)
  Evening 2-hour Postmeal: number analyzed (Participants) | 190 | 171
  Evening 2-hour Postmeal | 6.3 (3.36) | 12.2 (3.54)
  Bedtime: number analyzed (Participants) | 180 | 169
  Bedtime | 8.6 (6.37) | 19.0 (6.58)

9. Secondary Outcome: Change From Baseline in Insulin Dose at Week 16
Description: LS mean was determined by MMRM model with covariates: Baseline + Pooled Country + + Hemoglobin A1C Stratum + Personal CGM or FGM use during study flag + Treatment + Time + Treatment*Time (Type III sum of squares). The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least one post-baseline basal insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units per day (U/day)
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 199 | 186
units per day (U/day)
  Daily Basal Insulin Dose | -0.2 (0.43) | -0.1 (0.44)
  Daily Bolus Insulin Dose: number analyzed (Participants) | 197 | 183
  Daily Bolus Insulin Dose | 0.8 (0.66) | -1.0 (0.68)
  Total Daily Insulin Dose: number analyzed (Participants) | 195 | 183
  Total Daily Insulin Dose | 0.6 (0.80) | -1.1 (0.82)

10. Secondary Outcome: Change From Baseline in Bolus/Total Insulin Dose Ratio at Week 16
Description: The bolus/total ratio was derived as the bolus dose divided by the total insulin dose at each visit. LS mean was determined by MMRM model with covariates: Baseline + Pooled Country + + Hemoglobin A1C Stratum + Personal CGM or FGM use during study flag + Treatment + Time + Treatment*Time (Type III sum of squares). The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 16
Population: All randomized participants with non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: Percentage of bolus/total insulin dose
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 195 | 183
Percentage of bolus/total insulin dose | 0.6 (0.66) | -1.3 (0.68)

11. Secondary Outcome: Percentage of Participants With HbA1c <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 16
Population: All randomized participants with baseline and at least one post-baseline HbA1c <7% data. Missing endpoints were imputed by applying the Last Observation Carried Forward (LOCF) method to the post-baseline data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 207 | 191
Percentage of participants | 20.77 | 18.85

12. Secondary Outcome: Percentage of Participants With at Least 1 Pump Occlusion Alarm That Leads to an Unplanned Infusion Set Change
Description: Percentage of participants with at least 1 pump occlusion alarm that leads to an unplanned infusion set change was evaluated.
Time Frame: Baseline through Week 16
Population: All randomized participants with baseline and at least one post-baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 212 | 210
Percentage of participants | 12.7 | 14.8

13. Secondary Outcome: Percentage of Participants With at Least 1 Event of Unexplained Hyperglycemia >300 mg/dL Confirmed by SMBG That Leads to an Unplanned Infusion Set Change
Description: Percentage of participants with at least 1 event of unexplained hyperglycemia >300 milligrams per deciliter (mg/dL) confirmed by SMBG that leads to an unplanned infusion set change was evaluated.
Time Frame: Baseline through Week 16
Population: All randomized participants with baseline and at least one post-baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
Number analyzed (Participants) | 217 | 215
Percentage of participants | 18.4 | 16.3

ADVERSE EVENTS:
Time Frame: Up to 20 Weeks
Description: All randomized participants. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Insulin Lispro (Humalog) Lead-in; Insulin Lispro (Humalog): Participants received individual dose of 100 U/mL insulin lispro (Humalog) by CSII; where mealtime boluses were delivered 0 to 2 minutes prior to the start of each meal, with basal infusion rates 24 hours/day, and correction boluses as necessary.
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | Ultra-Rapid Lispro
All-Cause Mortality (participants affected / at risk) | 0/471 | 0/217 | 0/215
Serious Adverse Events (participants affected / at risk) | 4/471 | 10/217 | 17/215
Other Adverse Events (participants affected / at risk) | 15/471 | 31/217 | 90/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=471) | Insulin Lispro (Humalog) (N=217) | Ultra-Rapid Lispro (N=215)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/261 (0) | 1/119 (1) | 0/120 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 5 (6)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=471) | Insulin Lispro (Humalog) (N=217) | Ultra-Rapid Lispro (N=215)
Infusion site pain (General disorders) | 3 (3) | 6 (6) | 35 (41)
Infusion site reaction (General disorders) | 6 (6) | 16 (16) | 47 (60)
Nasopharyngitis (Infections and infestations) | 6 (6) | 13 (14) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03830281/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT03830281/SAP_001.pdf